CLINICAL TRIAL: NCT03448900
Title: Intervention Study for Smoking Cessation in Spanish College Students: Pragmatic Randomized Controlled Trial
Brief Title: Intervention Study for Smoking Cessation in Spanish College Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Collaborators: University of Navarra (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Smoking
Record Dates: First submitted 2018-02-20; First posted 2018-02-28 (Actual); Last update posted 2018-03-01 (Actual); Status verified 2018-02

CONDITIONS: Smoking; Smoking Cessation
Keywords: Cessation; College student; Motivational Interview; Self-efficacy; Intention; Beliefs; Young adult
MeSH Terms: conditions — Smoking; Smoking Cessation | interventions — Crisis Intervention

STUDY DESIGN:
Who Masked: Participant
Masking Description: Randomization was performed by one member of the research team who generated a blocked random number sequence, using EpiInfo version 7.0.9.7, and prepared the sealed opaque sequentially numbered envelopes (1-255) with the corresponding condition written inside. After each student agreed to participate in the study, the enve- lope was opened, determining the group to which he or she would be assigned. Students were unaware of the group assignments and randomization scheme.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multicomponent intervention (Experimental): The intervention group consisted in face-to-face 50-minute meeting [motivational interviewing (MI)]; online self-help material focused on: (1) decisions; (2) moods; (3) social life; (4) smoking health effects; and (5) quitting; e-mail 15 days before the MI, group therapy 2 months after the MI (60 minutes), a second follow-up visit 4 months after the MI (20 minutes).
  Interventions: Behavioral: Multicomponent intervention
- Brief advice (Active Comparator): The control group received a brief advice (5-10minutes) and a self-help pamphlet called 'Stop smoking'. Before giving brief advice, the nurse assessed smokers' habits and their willingness to quit. As is usually in this type of studies there were no follow-up sessions for this group.
  Interventions: Behavioral: Brief advice

INTERVENTIONS:
Behavioral: Multicomponent intervention — Motivational interview (50 minutes), on-line self-help material, support e-mail, group therapy, and second motivational interview (20 minutes)
  Arms: Multicomponent intervention
Behavioral: Brief advice — Brief advice (5-10minutes) and a self-help pamphlet
  Arms: Brief advice

SUMMARY:
This study evaluate the effectiveness of a nurse multi-component intervention aimed at helping Spanish college student smokers to quit smoking.

DETAILED DESCRIPTION:
This study hipotetize that a multicomponent intervention, tailored to college student and conducted by a nurse is more effective than brief advise.

The intervention was a multi-component intervention based on the Theory of Triadic Influence and on previous recommendations made in the Surgeon General's report . The strategies of this program consisted of a 50-minute motivational interview conducted by a nurse and online self-help material. The follow-up included a reinforcing e-mail and group therapy. The smoking-related Self-efficacy, Belief and Intention scale was used to assess outcomes.

ELIGIBILITY:
Inclusion Criteria

- Undergraduate or master students that smoked an average of at least one cigarette a week within the last 6 months

Exclusion Criteria

- Students who are ex-smokers

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 255 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2014-05 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Smoking cessation | 6 month follow-up
  The difference in the proportion of students who stopped smoking, between intervention and control subjects.

SECONDARY OUTCOMES:
Mean of smoked cigaretes | 6 month follow-up
  Among students that continued smoking the difference in the mean of cigarrete per day between intervention and control subjects; the difference in the mean of this variable pre- and post-intervention or control program
Quit attempts | 6 month follow-up
  Among students that continued smoking the difference in the numbers of quit attempts between intervention and control subjects
Stages of change according to Prochaska's model | 6 month follow-up
  The difference in the distribution on the stages of change between intervention and control subjects at 6 month follow-up
The self-efficacy to avoid smoking, and | 6 month follow-up
  the difference in the mean of self-efficacy to avoid smoking between intervention and control subjects; the difference in the mean of this variable pre- and post-intervention or control program; and the proportion of the total effect of smoking cessation explained by self-efficacy to avoid smoking.
Smoking-related beliefs | 6 month follow-up
  the difference in the mean of smoking-related beliefs between intervention and control subjects; the difference in the mean of this variable pre- and post-intervention or control program; and the proportion of the total effect of smoking cessation explained by smoking-related beliefs.
Intention to quit smoking | 6 month follow-up
  the difference in the mean of intention to quit smoking between intervention and control subjects; the difference in the mean of this variable pre- and post-intervention or control program; and the proportion of the total effect of smoking cessation explained by intention to stop smoking.

CONTACTS AND LOCATIONS:
Overall Officials: Miren I Pardavila-Belio, PhD, Principal Investigator — University of Navarra
Locations (1):
- Miren Idoia Pardavila Belio, Pamplona, Navarre, Spain

REFERENCES:
- [Result] Pardavila-Belio MI, Garcia-Vivar C, Pimenta AM, Canga-Armayor A, Pueyo-Garrigues S, Canga-Armayor N. Intervention study for smoking cessation in Spanish college students: pragmatic randomized controlled trial. Addiction. 2015 Oct;110(10):1676-83. doi: 10.1111/add.13009. Epub 2015 Jul 2. PMID 26053958
- [Result] Pardavila-Belio MI, Canga-Armayor A, Duaso MJ, Pueyo-Garrigues S, Pueyo-Garrigues M, Canga-Armayor N. Understanding how a smoking cessation intervention changes beliefs, self-efficacy, and intention to quit: a secondary analysis of a pragmatic randomized controlled trial. Transl Behav Med. 2019 Jan 1;9(1):58-66. doi: 10.1093/tbm/ibx070. PMID 30590861